CLINICAL TRIAL: NCT00808340
Title: Comparison of Three Soft Bifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-1485FA
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Results first posted 2010-08-26 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant

ARMS (6):
- senofilA test/senofilA prod/balafilconA (Active Comparator): Subjects wear 3 multifocal contact lenses: senofilcon A test worn first, senofilcon A production worn second, and balafilcon A worn third.
  Interventions: Device: balafilcon A; Device: senofilcon A production; Device: senofilcon A test
- senofilcon A test/balafilcon A/senofilcon A prod (Active Comparator): Subjects wear 3 multifocal contact lenses: senofilcon A test worn first, balafilcon A worn second, and senofilcon A production worn third.
  Interventions: Device: balafilcon A; Device: senofilcon A production; Device: senofilcon A test
- senofilcon A prod/senofilcon A test/balafilcon A (Active Comparator): Subjects wear 3 multifocal contact lenses: senofilcon A production worn first, senofilcon A test worn second, and balafilcon A worn third.
  Interventions: Device: balafilcon A; Device: senofilcon A production; Device: senofilcon A test
- senofilcon A prod/ balifilcon A/ senofilcon A test (Active Comparator): Subjects wear 3 multifocal contact lenses: senofilcon A production worn first, balafilcon A worn second, and senofilcon A test worn third.
  Interventions: Device: balafilcon A; Device: senofilcon A production; Device: senofilcon A test
- balafilcon A/senofilcon A test/senofilcon A prod (Active Comparator): Subjects wear 3 multifocal contact lenses: balafilcon A worn first, senofilcon A test worn second, and senofilcon A production worn third.
  Interventions: Device: balafilcon A; Device: senofilcon A production; Device: senofilcon A test
- balafilcon A/senofilcon A prod/senofilcon A test (Active Comparator): Subjects wear 3 multifocal contact lenses: balafilcon A worn first, senofilcon A production worn second, senofilcon A test worn third.
  Interventions: Device: balafilcon A; Device: senofilcon A production; Device: senofilcon A test

INTERVENTIONS:
Device: balafilcon A — multifocal contact lens
Device: senofilcon A production — multifocal contact lens
Device: senofilcon A test — multifocal contact lens

SUMMARY:
The primary purpose of the study is to compare the performance of three soft bifocal contact lenses in terms of the vision provided by the lenses.

ELIGIBILITY:
Inclusion Criteria:

* The subject must between 35 and 70 years of age.
* The subject must respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" or be already wearing presbyopic contact lens correction ( e.g. reading spectacles over contact lenses, multifocal or monovision contact lenses etc.).
* The subject's spherical equivalent distance refraction must be in the range of -1.00 to -6.00 in each eye.
* Refractive cylinder must be less than or equal to -0.75 D in each eye.
* The subject must have an add power of +0.75D to +2.50D in each eye.
* The subject must have best corrected visual acuity of 20/20-3 or better in each eye.
* The subject's must have at least 20/30-distance vision with the study contact lenses.
* The subject must agree that they are comfortable with their vision prior to being dispensed the study lenses.
* The subject must be an adapted soft contact lens wearer in both eyes.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must read and sign the STATEMENT OF INFORMED CONSENT and be provided a copy of the form.

Exclusion Criteria:

* Ocular or systemic allergies or disease that may interfere with contact lens wear.
* Systemic disease, autoimmune disease or use of medication, which may interfere with contact lens wear.
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining or any other abnormality of the cornea, which may contraindicate contact lens wear.
* Clinically significant (grade 3 or 4) tarsal abnormalities that might interfere with contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Pregnancy or lactation
* Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV).
* History of diabetes. History of binocular vision abnormality or strabismus.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2008-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Roanoke, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Senofilcon A Test/Senofilcon A Prod/Balafilcon A: Subjects wear 3 multifocal contact lenses: senofilcon A test worn first, senofilcon A production worn second, and balafilcon A worn third.
- Senofilcon A Prod/Senofilcon A Test/Balafilcon A: Subjects wear 3 multifocal contact lenses: senofilcon A prod worn first, senofilcon A test worn second, and balafilcon A worn third.
- Senofilcon A Prod/ Balifilcon A/ Senofilcon A Test: Subjects wear 3 multifocal contact lenses: senofilcon A prod worn first, balafilcon A worn second, and senofilcon A test worn third.
- Balafilcon A/Senofilcon A Prod/Senofilcon A Test: Subjects wear 3 multifocal contact lenses: balafilcon A worn first, senofilcon A producton worn second, senofilcon A test worn third.
Period: First Intervention
Arm/Group | Senofilcon A Test/Senofilcon A Prod/Balafilcon A | Senofilcon A Test/Balafilcon A/Senofilcon A Prod | Senofilcon A Prod/Senofilcon A Test/Balafilcon A | Senofilcon A Prod/ Balifilcon A/ Senofilcon A Test | Balafilcon A/Senofilcon A Test/Senofilcon A Prod | Balafilcon A/Senofilcon A Prod/Senofilcon A Test
Started | 4 | 9 | 7 | 3 | 5 | 6
Completed | 4 | 9 | 7 | 3 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Senofilcon A Test/Senofilcon A Prod/Balafilcon A | Senofilcon A Test/Balafilcon A/Senofilcon A Prod | Senofilcon A Prod/Senofilcon A Test/Balafilcon A | Senofilcon A Prod/ Balifilcon A/ Senofilcon A Test | Balafilcon A/Senofilcon A Test/Senofilcon A Prod | Balafilcon A/Senofilcon A Prod/Senofilcon A Test
Started | 4 | 9 | 7 | 3 | 5 | 6
Completed | 4 | 9 | 7 | 3 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Senofilcon A Test/Senofilcon A Prod/Balafilcon A | Senofilcon A Test/Balafilcon A/Senofilcon A Prod | Senofilcon A Prod/Senofilcon A Test/Balafilcon A | Senofilcon A Prod/ Balifilcon A/ Senofilcon A Test | Balafilcon A/Senofilcon A Test/Senofilcon A Prod | Balafilcon A/Senofilcon A Prod/Senofilcon A Test
Started | 4 | 9 | 7 | 3 | 5 | 6
Completed | 4 | 9 | 7 | 3 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] — Overall completed study population
  years | 50.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Distance Bright Illumination Binocular Visual Performance Reported as Visual Acuity
Description: Tested with both eyes together in bright lighting, reading charts distant to the subject. This outcome is measured in logMAR units.LogMAR stands for the logarithm of the minimum angle of resolution. Ideal is 0.0 and represents 20/20 Snellen acuity. logMAR values > 0.00 indicate vision poorer than the ideal and values <0.00 indicate vision greater than the ideal.
Time Frame: 5 minutes after insertion
Measure: Least Squares Mean (Standard Error); unit: logMAR
Groups:
- Senofilcon A Test: senofilcon A test represents subjects that wore this lens in either the first, second, or third period.
- Senofilcon A Prod: senofilcon A prod represents subjects that wore this lens in either the first, second, or third period.
- Balafilcon A: balafilcon A represents subjects that wore this lens in either the first, second, or third period.
Arm/Group | Senofilcon A Test | Senofilcon A Prod | Balafilcon A
Number analyzed (Participants) | 34 | 34 | 34
logMAR | 0.8191 (0.161) | 0.6942 (0.161) | 1.0635 (0.161)
Statistical Analysis 1: Comparison: Senofilcon A Test vs Senofilcon A Prod; Alternative hypothesis is that senofilcon A multifocal prod is non-inferior to senofilcon A multifocal test; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.1249, 97.5% CI 2-sided [-0.4143 to 0.1644], Standard Error of Mean 0.1464 — Mean difference is calculated as senofilcon A multifocal prod minus senofilcon A multifocal test
Statistical Analysis 2: Comparison: Senofilcon A Prod vs Balafilcon A; Alternative hypothesis is that senofilcon A multifocal prod is non-inferior to balafilcon A multifocal; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.3693, 97.5% CI 2-sided [-0.6587 to -0.07996], Standard Error of Mean 0.1464 — The mean difference was calculated as balafilcon A multifocal minus senofilcon A multifocal prod

2. Primary Outcome: Near Bright Illumination Binocular Visual Performance Reported as Visual Acuity
Description: Tested with both eyes together in bright lighting reading charts near to the subject. This outcome is measured in logMAR units.LogMAR stands for the logarithm of the minimum angle of resolution. Ideal is 0.0 and represents 20/20 Snellen acuity. logMAR values > 0.00 indicate vision poorer than the ideal and values <0.00 indicate vision greater than the ideal.
Time Frame: 5 minutes after insertion
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | Senofilcon A Test | Senofilcon A Prod | Balafilcon A
Number analyzed (Participants) | 34 | 34 | 34
logMAR | -0.6735 (0.161) | -0.6327 (0.161) | -0.1719 (0.161)
Statistical Analysis 1: Comparison: Senofilcon A Test vs Senofilcon A Prod; Alternative hypothesis is that senofilcon A multifocal prod is non-inferior to senofilcon A multifocal test; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.04083, 97.5% CI 2-sided [-0.2485 to 0.3302], Standard Error of Mean 0.1464 — The mean difference is calculated as senofilcon A multifocal prod minus senofilcon A multifocal test
Statistical Analysis 2: Comparison: Senofilcon A Prod vs Balafilcon A; Alternative hypothesis is that senofilcon A multifocal prod is non-inferior to balafilcon A multifocal; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.4608, 97.5% CI 2-sided [-0.7502 to -0.1714], Standard Error of Mean 0.1464 — The mean difference was calculated as senofilcon A multifocal prod minus balafilcon A multifocal

3. Primary Outcome: Type of Corneal Staining
Description: Investigator rated type of corneal staining as either 0=none, 1=micropunctate, 2=macropunctate, 3=coalesced, or 4=patch(> or = to mm).
Time Frame: after 1 week of lens wear, for each lens type
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A Test | Senofilcon A Prod | Balafilcon A
Number analyzed (Participants) | 34 | 34 | 34
Units on a scale | 0.1311 (0.07154) | 0.1017 (0.07154) | 0.1694 (0.07154)
Statistical Analysis 1: Comparison: Senofilcon A Test vs Senofilcon A Prod; Alternative hypothesis is senofilcon A multifocal prod is non-inferior to senofilcon A multifocal test; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.02941, 97.5% CI 2-sided [-0.08153 to 0.02271], Standard Error of Mean 0.02656 — The mean difference is calculated as senofilcon A multifocal prod minus senofilcon A multifocal test
Statistical Analysis 2: Comparison: Senofilcon A Prod vs Balafilcon A; Alternative hypothesis is senofilcon A multifocal prod is non-inferior to balafilcon A multifocal; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.06765, 97.5% CI 2-sided [-0.1198 to -0.01553], Standard Error of Mean 0.02656 — The mean difference is calculated as senfilcon A multifocal prod minus balafilcon A multifocal

4. Primary Outcome: Overall Subjective Vision
Description: Subject rated the overall quality of vision with the study contact lenses. 5=excellent, 4=very good, 3=good, 2=fair, 1=poor.
Time Frame: after 1 week of lens wear, for each lens type
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A Test | Senofilcon A Prod | Balafilcon A
Number analyzed (Participants) | 34 | 34 | 34
Units on a scale | 3.5373 (0.1681) | 3.207 (0.1681) | 3.4351 (0.1681)
Statistical Analysis 1: Comparison: Senofilcon A Test vs Senofilcon A Prod; Alternative hyposthesis is that senofilcon A multifocal prod is non-inferior to senofilcon A multifocal test; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.3304, 97.5% CI 2-sided [-0.779 to 0.1183], Standard Error of Mean 0.2243 — The mean difference is calculated as senofilcon A multifocal prod minus senofilcon A multifocal test
Statistical Analysis 2: Comparison: Senofilcon A Prod vs Balafilcon A; Alternativie hypothesis is that senofilcon A multifocal prod is non-inferior to balafilcon A multifocal; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.2281, 97.5% CI 2-sided [-0.6767 to 0.2206], Standard Error of Mean 0.2243 — The mean difference is calculated as senofilcon A multifocal prod minus balafilcon A multifocal

ADVERSE EVENTS:
Arm/Group | Senofilcon A Test | Senofilcon A Prod | Balafilcon A
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.